CLINICAL TRIAL: NCT01593163
Title: Randomised Controlled Clinical Trial of Echocardiographically Guided Versus Standard Ibuprofen Treatment for Patent Ductus Arteriosus: a Pilot Study
Brief Title: Echocardiographically Guided Versus Standard Ibuprofen Treatment for Patent Ductus Arteriosus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario la Paz (Other)
Responsible Party: Principal Investigator, Maria Carmen Bravo Laguna, Principal Investigator, Fundacion para la Investigacion Biomedica del Hospital Universitario la Paz
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IbuEchoG
Record Dates: First submitted 2012-05-03; First posted 2012-05-08 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Patent Ductus Arteriosus
Keywords: Functional echocardiography; power Doppler cranial ultrasonography; N-terminal probrain natriuretic peptide; Patent ductus arteriosus
MeSH Terms: conditions — Ductus Arteriosus, Patent

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EchoG (Experimental): Infants in the experimental group (echoG treatment) received additional doses of ibuprofen only if PDA was still ≥ 1.5 mm at the time of the corresponding ibuprofen dose.
  Interventions: Drug: Ibuprofen EchoG
- ST (standard treatment) (Other): Infants received 3 doses of ibuprofen at 24-hour intervals, independently of ductal size, as long as additional doses were not contraindicated.
  Interventions: Drug: Standard ibuprofen treatment

INTERVENTIONS:
Drug: Ibuprofen EchoG — Infants in the experimental group (echoG treatment) received additional doses of ibuprofen only if PDA was still ≥ 1.5 mm at the time of the corresponding ibuprofen dose.
  Other Names: Echocardiographically guided ibuprofen treatment
  Arms: EchoG
Drug: Standard ibuprofen treatment — Infants received 3 doses of ibuprofen at 24-hour intervals, independently of ductal size, as long as additional doses were not contraindicated.
  Arms: ST (standard treatment)

SUMMARY:
Patent ductus arteriosus (PDA) is a very common condition in immature newborn babies and it has been associated to morbidity and mortality. Ibuprofen is the drug of choice for PDA treatment according to the last version of the Cochrane review. Nowadays the best dose regimen for ibuprofen remains uncertain. The investigators aim to perform a randomized controlled clinical trial to assess whether echocardiographically guided PDA ibuprofen treatment versus standard treatment could reduce the number of doses of ibuprofen without increasing the reopening rate and reducing the side effects associated to this medication.

DETAILED DESCRIPTION:
Patent ductus arteriosus (PDA) is presented in 55 to 70% of the preterm infants with a gestational age lower than 30 weeks or a birth weight lower than 1000 grams. PDA has being associated to mortality or morbidity such as ischemic or hemorrhagic cerebral events, necrotising enterocolitis, renal disfunction or poor pulmonary outcome; however, it is not clear whether these are a consequence of the PDA presence, the treatment implemented for closing it, or the immaturity of these population. PDA standard treatment (ST) consists on three doses of indomethacin or ibuprofen (10-5-5mg/kg) given 24 hours apart, being the surgical closure a second line therapeutic option. In spite of ibuprofen has been pointed as the drug of choice for PDA treatment by the last version of the Cochrane review, side effects have been associated to both medication. Standard ibuprofen treatment is based on a clinical trial where the three-dose protocol seemed to be more effective than one-dose scheme for PDA closure; however, the sample size was not powered to find differences statistically significant, so nowadays the best dose regimen for ibuprofen remains uncertain. Functional echocardiographic assessment is spreading to all over the world. In this scenario, it has been proposed its implementation to guide PDA treatment in order to individualize the number of doses of indomethacin administered as a function of patient's response, limiting the doses and side effects in those where PDA presented an early constriction. The investigators hypothesized whether echocardiographically guided PDA ibuprofen treatment could reduce the number of doses of ibuprofen without increasing the reopening rate and reducing the side effects associated to this medication.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants with a gestational age lower than 37 weeks of gestational age
* PDA ≥ 1.5 mm
* No contraindication to receive ibuprofen
* Informed consent signed.

Exclusion Criteria:

* Life-threatening congenital defects
* Congenital heart disease
* Contraindication for ibuprofen administration such as oligoanuria < 1cc/kg/h or recent severe intraventricular bleeding (IVH grade III) or creatinine serum level > 1.5 mg/dl or potential intestinal ischemia.
* Informed consent refused

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2009-05; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
PDA re-opening rate | Infants will be followed for the duration of hospital stay in the Newborn Unit, an expected average of 4-8 weeks
  PDA re-opening after echocardiographically documented closure, which the attending physician deemed amenable to additional treatment. Infants with ventilator weaning difficulty, protracted metabolic acidosis or persistent hemodynamic instability were included in this category.

SECONDARY OUTCOMES:
treatment failure | Infants will be followed for the duration of hospital stay in the Newborn Unit, an expected average of 4-8 weeks
  PDA ≥ 1.5 mm 24 hours after a complete ibuprofen course
need for surgical ligation | Infants will be followed for the duration of hospital stay in the Newborn Unit, an expected average of 4-8 weeks
  need for surgical ligation
need for additional ibuprofen doses | Infants will be followed for the duration of hospital stay in the Newborn Unit, an expected average of 4-8 weeks
  need for additional ibuprofen doses after treatment was completed
urine output | before the first ibuprofen dose was administered (between 12-72 hours of life) until 24 hours after the last dose of ibuprofen was administered (between 36-168 h of life)
  urine output
serum creatinine | before the first ibuprofen dose was administered (between 12-72 hours of life) until 24 hours after the last dose of ibuprofen was administered (between 36-168 h of life)
  serum creatinine
mortality | Infants will be followed for the duration of hospital stay in the Newborn Unit, an expected average of 4-8 weeks
  mortality
bronchopulmonary dysplasia | Infants will be followed for the duration of hospital stay in the Newborn Unit, an expected average of 4-8 weeks
  bronchopulmonary dysplasia (O2 need at 36 postmenstrual weeks)
necrotising enterocolitis | Infants will be followed for the duration of hospital stay in the Newborn Unit, an expected average of 4-8 weeks
  necrotising enterocolitis
intraventricular hemorrhage | Infants will be followed for the duration of hospital stay in the Newborn Unit, an expected average of 4-8 weeks
  intraventricular hemorrhage
White matter damage | Infants will be followed for the duration of hospital stay in the Newborn Unit, an expected average of 4-8 weeks
  White matter damage
Laser therapy for retinopathy | Infants will be followed for the duration of hospital stay in the Newborn Unit, an expected average of 4-8 weeks
  Laser therapy for retinopathy
peak systolic velocity | before each ibuprofen dose should be administered (3 days) and 24 hours after the last dose of ibuprofen was administered
  peak systolic velocity measured by means of cerebral Doppler ultrasonography in the anterior and middle cerebral arteries
end-diastolic velocity | before each ibuprofen dose should be administered (3 days) and 24 hours after the last dose of ibuprofen was administered
  end-diastolic velocity measured by means of cerebral Doppler ultrasonography in the anterior and middle cerebral arteries
resistance index | before each ibuprofen dose should be administered (3 days) and 24 hours after the last dose of ibuprofen was administered
  resistance index measured by means of cerebral Doppler ultrasonography in the anterior and middle cerebral arteries
pulsatility index | before each ibuprofen dose should be administered (3 days) and 24 hours after the last dose of ibuprofen was administered
  pulsatility index measured by means of cerebral Doppler ultrasonography in the anterior and middle cerebral arteries

CONTACTS AND LOCATIONS:
Overall Officials: María Carmen Bravo, PhD MD, Principal Investigator — Department of Neonatology, La Paz University Hospital; Fernando Cabañas, PhDMD, Study Chair — Department of Neonatology, La Paz University Hospital; Joan Riera, Bio-Engineer, Study Chair — Department of Neonatology, La Paz University Hospital; Elia Pérez-Fernández, Study Chair — Division of Statistics, La Paz University Hospital. Madrid, Spain.; José Quero, PhDMD, Study Chair — Department of Neonatology, La Paz University Hospital. Madrid, Spain.; Jesús Pérez-Rodríguez, PhDMD, Study Chair — Department of Neonatology, La Paz University Hospital. Madrid, Spain.; Adelina Pellicer, PhDMD, Study Director — Department of Neonatology, La Paz University Hospital. Madrid, Spain.
Locations (1):
- Department of Neonatology, La Paz University Hospital, Madrid, Madrid, Spain

REFERENCES:
- [Background] Carmo KB, Evans N, Paradisis M. Duration of indomethacin treatment of the preterm patent ductus arteriosus as directed by echocardiography. J Pediatr. 2009 Dec;155(6):819-822.e1. doi: 10.1016/j.jpeds.2009.06.013. Epub 2009 Jul 29. PMID 19643435